CLINICAL TRIAL: NCT07345715
Title: Comparison Between Oral Melatonin Versus Nebulized Dexmedetomidine on Emergence Agitation in Children Undergoing Adenotonsillectomy: A Prospective, Randomized Controlled Trial
Brief Title: Oral Melatonin Versus Nebulized Dexmedetomidine on Emergence Agitation in Children Undergoing Adenotonsillectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Abd Elsamd Kamel Eid, Assistant Lecturer of Anesthesia, Surgical Intensive Care and Pain Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD430/6/25
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Oral Melatonin; Nebulized Dexmedetomidine; Emergence Agitation; Children; Adenotonsillectomy
MeSH Terms: conditions — Emergence Delirium | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group C (Control Group) (Active Comparator): Participants will receive placebo nebulizer (3 ml of normal saline) without drug and 0.5 mg/kg of midazolam dissolved in Apple Juice.
  Interventions: Drug: Normal saline
- Melatonin Group (Experimental): Participants will receive placebo nebulizer (3 ml of normal saline) without drug and 0.2 mg/kg of oral melatonin syrup.
  Interventions: Drug: Oral melatonin syrup
- Dexmedetomidine Group (Experimental): Participants will receive placebo syrup (Apple Juice) and 2 µ/kg nebulized dexmedetomidine prepared in 0.9% normal saline to a final volume of 3ml.
  Interventions: Drug: Nebulized dexmedetomidine

INTERVENTIONS:
Drug: Normal saline — Participants will receive placebo nebulizer (3 ml of normal saline) without drug and 0.5 mg/kg of midazolam dissolved in Apple Juice.
  Arms: Group C (Control Group)
Drug: Oral melatonin syrup — Participants will receive placebo nebulizer (3 ml of normal saline) without drug and 0.2 mg/kg of oral melatonin syrup.
  Arms: Melatonin Group
Drug: Nebulized dexmedetomidine — Participants will receive placebo syrup (Apple Juice) and 2 µ/kg nebulized dexmedetomidine prepared in 0.9% normal saline to a final volume of 3ml.
  Arms: Dexmedetomidine Group

SUMMARY:
This study aims to compare the efficacy of using oral Melatonin versus nebulized Dexmedetomidine in limitation of emergence agitation in children undergoing adenotonsillectomy.

DETAILED DESCRIPTION:
Adenotonsillectomy is one of the most commonly performed surgical procedures in children with high incidence of emergence agitation about 80% and high degree of post operative pain.

Oral midazolam, a short-acting benzodiazepine, is commonly used as a standard premedication in children due to its well-established anxiolytic, sedative, and amnestic effects. It works by enhancing GABAergic neurotransmission in the central nervous system, helping reduce anxiety and facilitating a smoother anesthetic induction and emergence.

Dexmedetomidine is a centrally acting α-2 adrenergic agonist with sedative, hypnotic, analgesic, anxiolytic, anti-sialagogue, antinociceptive and sympatholytic action.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 3 and 7 years.
* Both sexes.
* Classified as American Society of Anesthesiologists (ASA) physical status I or II according to the American Society of Anesthesiologists.
* Scheduled for elective adenotonsillectomy under general anesthesia.

Exclusion Criteria:

* Parental refusal to participate in the study.
* Known allergy or hypersensitivity to dexmedetomidine, melatonin or midazolam.
* Presence of developmental delay.
* Central nervous system disorders.
* Intellectual disability (formerly termed mental retardation).
* Neurological or psychiatric conditions associated with anxiety or agitation (e.g., cerebral palsy, epilepsy, separation anxiety disorder, attention-deficit/hyperactivity disorder).
* Current or recent treatment with anticonvulsants or sedative medications

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Emergence agitation | 30 minutes after recovery
  Emergence agitation will be assessed by using Pediatric Anesthesia Emergence Delirium Scale (PAED). The PAED scale consists of 5 criteria that are scored using a 5-point scale. The scores of each criterion are added to make a total score. The maximum achievable score is 20. A score of ≥10 has 64% sensitivity and 86% specificity for the diagnosis of Emergence Agitation (ED). A score of >12 has 100% sensitivity and 94.5% specificity for the diagnosis of ED.

SECONDARY OUTCOMES:
Perioperative anxiety | During transferring to operating room (Up to 30 minutes).
  Perioperative anxiety which will be measured by using Parental separation anxiety scale (PSAS).
  PSAS scale:
  1. Excellent: Patient unafraid, cooperative, or asleep.
  2. Good: Slight fear and or crying, quiet with reassurance.
  3. Fair: Moderate fear and crying, not quiet with reassurance.
  4. Poor: Crying, need for restraint. Score of 1 or 2 were classified as an acceptable separation, whereas scores of 3 or 4 were considered difficult separations from the parents.
Mask tolerance | Intraoperatively
  Mask tolerance which will be measured by using mask acceptance scale (MAS).
  MAS score:
  1. Excellent: calm, cooperative, or asleep.
  2. Good: Moderate fear of the mask Manageable with reassurance.
  3. Fair: Cries, combative and needs restraining.
  4. Poor: Crying, need for restraint. Score of 1 or 2 were classified as an acceptable mask tolerance, whereas scores of 3 or 4 were considered poor mask tolerance.
Degree of pain | Before home discharge (Up to 6 hours)
  Postoperative pain control will be assessed using Face, Legs, Activity, Cry, Consolability (FLACC) ) on arrival to PACU, 30 minutes, one hour, two hours after surgery and before home discharge.
  Each category is scored on the 0-2 scale, which results in a total score of 0-10.
  * 0 = Relaxed and comfortable.
  * 1-3 = Mild discomfort.
  * 4-6 = Moderate pain.
  * 7-10 = Severe discomfort/pain.
Total postoperative analgesics consumption | Before home discharge (Up to 6 hours)
  Total postoperative analgesics consumption will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.